CLINICAL TRIAL: NCT03317041
Title: Effects of a Capacitive-resistive Electric Transfer Therapy Exposure on Physiological and Biomechanical Parameters in Recreational Runners: a Randomized Controlled Crossover Trial
Brief Title: Capacitive-resistive Electric Transfer Therapy for Recovery From Running Fatigue
Acronym: UPV/EHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Iraia Bidaurrazaga-Letona, PhD, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 313-2015
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Running; Fatigue
Keywords: Capacitive-resistive electric transfer therapy; Radiofrequency therapy; Recovery intervention; Fatigue; Running
MeSH Terms: conditions — Fatigue | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecar treatment group (Experimental): The capacitive-resistive electric transfer (Tecar) therapy treatment group will receive 45 minutes of Tecar therapy treatment.
  Interventions: Other: Capacitive-resistive electric transfer (Tecar) therapy
- Control group (No Intervention): Participants will test passively in a sitting position for 30-min period

INTERVENTIONS:
Other: Capacitive-resistive electric transfer (Tecar) therapy — The Tecar treatment group will receive 45 minutes of Tecar therapy treatment. Subjects will lay down with the face down and two metallic plaques situated under each quadriceps muscle all over all the treatment. The treatment will start with the automatic capacitive energy transfer for 10-min where the capacitive plaque is situated on the sole of each foot with an elastic band. After that, the capacitive plaque will be pulled out. Then, the resistive electrode will be moved longitudinally through different muscles with massage lotion during 15-min per each lower extremity. The treatment will conclude with the automatic capacitive energy transfer for 10-min and the capacitive plaque situated on the sole of each foot with an elastic band.
  Arms: Tecar treatment group

SUMMARY:
Reducing fatigue and improving the recovery capabilities of runners has gained more interest over the last years. Recently, capacitive-resistive electric transfer (Tecar) therapy is commonly used by physical therapists to help athletes recover from muscle fatigue. However, empiric evidence supporting the benefits of Tecar to recovery is lacking. This study investigated the effects of a Tecar treatment performed shortly after an exhausting training session on both physiological and biomechanical parameters of running.

DETAILED DESCRIPTION:
In this randomized controlled crossover trial all subjects will perform two test protocols separated by 2 weeks. Each protocol will comprise one exhausting training session (20-min warm-up consisted of 15-min of continuous self-paced running followed by 5-min of fast-finish progression runs increasing speeds (from approximately 60% to 80% of maximal heart rate, participant controlled), 10 x 500 m sprints at 90% of maximal heart rate with a 2-min rest period between bouts and a recovery phase consisting of 10-min of slow jogging). Twenty-four hours after this exhausting training, subjects will perform an incremental running test on a treadmill (Pre-intervention test) where subjects will start at 10 km/h for 6 min after which speed will be increased by 2 km/h every 6 min until a 16 km/h trial is completed. One hour after this test, in one protocol subjects will receive Tecar therapy (Tecar treatment group); in the other group (Control group) participants will rest passively in a sitting position for 30-min period. To evaluate the relevance of the changes induced by Tecar therapy/passive recovery, subjects will repeat the treadmill test 48 hours after the first test in both groups (72 hours after the exhaustive training).

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (current participation in races and a 10-km race time <34.5-min)

Exclusion Criteria:

* Suffered from any injury within the preceding 4 months.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
CHANGE FROM BASELINE OXYGEN UPTAKE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Oxygen uptake (mL kg-1 min-1) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Oxygen uptake will be recorded using a gas analyzer system (Esgostik Geratherm, Geschwenda, Germany).
CHANGE FROM BASELINE RESPIRATORY EXCHANGE RATIO AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Respiratory exchange ratio (ratio between the amount of carbon dioxide (CO2) produced in metabolism and oxygen (O2)) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Respiratory exchange ratio will be recorded using a gas analyzer system (Esgostik Geratherm, Geschwenda, Germany).
CHANGE FROM BASELINE VENTILATION AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Ventilation (L• min-1) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Ventilatory output will be recorded using a gas analyzer system (Esgostik Geratherm, Geschwenda, Germany).
CHANGE FROM BASELINE HEART RATE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Heart rate (beat • min-1) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Heart rate will be recorded by a heart monitor (Polar RS800, Kempele, Finland).
CHANGE FROM BASELINE BLOOD LACTATE CONCENTRATION AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  - Blood lactate concentration (mmol •L-1) will be assessed in an incremental running test on a treadmill (HP Cosmos pulsar, Nussdorf-Traunstein, Germany). Capillary blood samples will be obtained in each test from the earlobe for the determination of blood lactate concentration by a portable lactate analyzer (Lactate, Arkray, KDK Corporation, Kyoto, Japan).
CHANGE FROM BASELINE STRIDE LENGTH AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride length (cm), defined as the length the treadmill belt moves from toe-off to initial ground contact in successive steps, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE STRIDE FREQUENCY AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride frequency, defined as the number of ground contact events per minute, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE STRIDE ANGLE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Stride angle (º), defined as the angle of the parable tangent derived from the theoretical arc traced by a foot during a stride and the ground, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE GROUND CONTACT TIME AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Ground contact time (s), defined as the time from when the foot contacts the ground to when the toes left the ground and was determined by the disruption of the infrared gates, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE SWING TIME AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  The swing time (s) corresponds to the time from foot flat to initial take-off. Swing time will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE CONTACT PHASE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  Contact phase (%), defined as the percentage of the ground contact time at which the different sub-phases of stance phase occur, will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE SUPPORT PHASE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  The support sub-phase (%) corresponds to the time from initial ground contact to foot flat.
  Support phase will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.
CHANGE FROM BASELINE PUSH-OFF PHASE AT 48 HOURS AFTER THE TREATMENT. | Participants will be assessed at baseline (24 hours after an exhaustive training session) and at 48 hours after the treatment.
  The push-off phase (%) corresponds to the time from initial take-off to toe-off.
  Push-off phase will be measured using an optical measurement system (Optojump-next, Microgate, Bolzano, Italy) placed at the treadmill belt level.

SECONDARY OUTCOMES:
Body height (cm) | Participants will be assessed at baseline (24 hours after an exhaustive training session).
  Body height will be measured using a stadiometer (Año Sayol, Barcelona, Spain) following the guidelines outlined by the International Society for the Advancement of Kinanthropometry.
Body weight (kg) | Participants will be assessed at baseline (24 hours after an exhaustive training session).
  Body weight will be measured using a balance (Año Sayol, Barcelona, Spain) following the guidelines outlined by the International Society for the Advancement of Kinanthropometry.

IPD SHARING:
Plan to Share IPD: No